CLINICAL TRIAL: NCT04381871
Title: Phase II ,III Randomized Double Blind Parallel Arms Clinical Trial of Potential Role of Gum Arabic ( Acacia Senegal) as Immunomodulatory Agent Among COVID 19 Patients in Sudan
Brief Title: Potential Role of Gum Arabic as Immunomodulatory Agent Among COVID 19 Patients
Acronym: GA&COVID19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Neelain University (Other)
Collaborators: University of Khartoum (Other)
Responsible Party: Principal Investigator, Lamis Kaddam, Dr.Lamis Kaddam, Al-Neelain University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GA& COVID19
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: COVID 19
Keywords: Gum Arabic; Immunomodulator
MeSH Terms: conditions — COVID-19 | interventions — Gum Arabic; Pectins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This arm will receive 100% natural Gum Arabic provided in a powder form in 30-grams-dose
  Interventions: Dietary Supplement: Acacia Senegal
- Control group (Placebo Comparator): This group will be provided with pectin powder provided as one-gram-dose
  Interventions: Dietary Supplement: Pectin

INTERVENTIONS:
Dietary Supplement: Acacia Senegal — Oral Digestion of Gum Arabic to be consumed early morning on daily basis for 4weeks
  Other Names: Gum Arabic
  Arms: Intervention Group
Dietary Supplement: Pectin — Oral Digestion of Pectin to be consumed early morning on daily basis for 12 weeks
  Arms: Control group

SUMMARY:
To study the efficacy of Gum Arabic as an immuno modulator and anti-inflammatory agent among COVID 19 seropositive patients..Half of participants will receive Gum Arabic and the other half will receive placebo

DETAILED DESCRIPTION:
Randomized placebo controlled trial including COVID 19 seropositive patients will be treated with 30 gram per day for 4 weeks, compared to placebo group treated for the same duration in positive COVID 19 patients.

Blood samples will be taken first at base line level, after two weeks and after the intervention after satisfying the inclusion and exclusion criteria. The main objective is to assess the effect of Gum Arabic (acacia Senegal) on immune system among COVID-19 patients. The outcome of this project understand SARS-CoV-2 immune response in COVID patients and the effect of Gum Arabic (Acacia Senegal) consumption to counteract progression of the disease

ELIGIBILITY:
Inclusion Criteria:

* COVID 19 infected as proved by real time PCR (polymerase chain reaction) .( newly diagnosed)

Exclusion Criteria:

* Intubated patients on parental treatment

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline score of Immune Response to end of the trial ( Time Frame: up to 4 weeks ) | 4 weeks
  Changes of the level of Tumor Necrosis Factor (TNF), interleukin IL8,IL6,IL10 from the baseline values
Mortality rate | from the date of assignment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to two months
  The percentage of deaths among COVID 19 patients received Gum Arabic compared to placebo

SECONDARY OUTCOMES:
Determine viral load in each patient | 4 weeks
  Change of viral load from Baseline

OTHER OUTCOMES:
clinical improvement and hospital discharge | from the date of assignment until the date of hospital discharge for the last assigned case, whichever comes first, assessed up to two months
  Time of discharge from hospital after full recovery

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa KM Nimeiri, MD, Study Chair — Al Neelain University, Faculty of Medicine; Moawia M Mukhtar, PhD, Study Director — University of Khartom , Institute of Endemic Diseases
Locations (2):
- Sudan (2):
  - Omdurman Teaching Hospital, Khartoum, Omdurman
  - Jabra Hospital,, Khartoum

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali NE, Kaddam LA, Alkarib SY, Kaballo BG, Khalid SA, Higawee A, AbdElhabib A, AlaaAldeen A, Phillips AO, Saeed AM. Gum Arabic (Acacia Senegal) Augmented Total Antioxidant Capacity and Reduced C-Reactive Protein among Haemodialysis Patients in Phase II Trial. Int J Nephrol. 2020 Apr 9;2020:7214673. doi: 10.1155/2020/7214673. eCollection 2020. PMID 32328307
- [Background] Kamal E, Kaddam LA, Dahawi M, Osman M, Salih MA, Alagib A, Saeed A. Gum Arabic Fibers Decreased Inflammatory Markers and Disease Severity Score among Rheumatoid Arthritis Patients, Phase II Trial. Int J Rheumatol. 2018 Jul 5;2018:4197537. doi: 10.1155/2018/4197537. eCollection 2018. PMID 30112005
- [Background] Pan L, Mu M, Yang P, Sun Y, Wang R, Yan J, Li P, Hu B, Wang J, Hu C, Jin Y, Niu X, Ping R, Du Y, Li T, Xu G, Hu Q, Tu L. Clinical Characteristics of COVID-19 Patients With Digestive Symptoms in Hubei, China: A Descriptive, Cross-Sectional, Multicenter Study. Am J Gastroenterol. 2020 May;115(5):766-773. doi: 10.14309/ajg.0000000000000620. PMID 32287140
- [Background] Ruscitti P, Berardicurti O, Iagnocco A, Giacomelli R. Cytokine storm syndrome in severe COVID-19. Autoimmun Rev. 2020 Jul;19(7):102562. doi: 10.1016/j.autrev.2020.102562. Epub 2020 May 3. No abstract available. PMID 32376400
- [Derived] Kaddam L, Babiker R, Ali S, Satti S, Ali N, Elamin M, Mukhtar M, Elnimeiri M, Saeed A. Potential Role of Acacia Senegal (Gum Arabic) as Immunomodulatory Agent among newly diagnosed COVID 19 Patients: A structured summary of a protocol for a randomised, controlled, clinical trial. Trials. 2020 Sep 5;21(1):766. doi: 10.1186/s13063-020-04707-2. PMID 32891160